CLINICAL TRIAL: NCT01752634
Title: A Phase III Randomized, Double-blind, Placebo-controlled Multicenter Study of Subcutaneous Secukinumab in Prefilled Syringes to Demonstrate the Efficacy at 24 Weeks and to Assess the Long Term Efficacy, Safety and Tolerability up to 5 Years in Patients With Active Psoriatic Arthritis
Brief Title: Efficacy at 24 Weeks With Long Term Safety, Tolerability and Efficacy up to 5 Years of Secukinumab in Patients of Active Psoriatic Arthritis
Acronym: FUTURE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457F2312; 2012-004439-22 (EudraCT Number)
Record Dates: First submitted 2012-10-23; First posted 2012-12-19 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis, PsA, ACR, CASPAR, PASDAS
MeSH Terms: conditions — Arthritis, Psoriatic; Salivary Gland Adenoma, Pleomorphic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Secukinumab (AIN457) 75 mg s.c. (Experimental): Secukinumab 75 mg at BSL, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4.
  Interventions: Drug: Secukinumab (AIN457)
- Secukinumab (AIN457) 150 mg s.c. (Experimental): Secukinumab 150 mg at BSL, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4.
  Interventions: Drug: Secukinumab (AIN457)
- Secukinumab (AIN457) 300 mg s.c. (Experimental): Secukinumab 300 mg at BSL, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4
  Interventions: Drug: Secukinumab (AIN457)
- Placebo s.c. (Placebo Comparator): Placebo at BSL, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4. Non-responder (assessed at Week 16) were re-randomized to receive AIN457 150mg or AIN457 300 mg starting at Week 16. Responder (assessed at Week 16) were re-randomized to receive AIN457 150mg or AIN457 300 mg starting at Week 24.
  Interventions: Drug: Secukinumab (AIN457); Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab (AIN457) — Secukinumab (AIN457)
Drug: Placebo — Placebo PFS for s.c. administration.
  Arms: Placebo s.c.

SUMMARY:
This study was to provide 24 - 52 week efficacy, safety and tolerability data to support the registration of the secukinumab (AIN457) prefilled syringe (PFS) for subcutaneous self administration in subjects with active PsA despite current or previous NSAID, DMARD and/or anti-TNFα therapy. An additional 4 years of long-term efficacy and safety data were collected during the post Week 52 period of the study.

DETAILED DESCRIPTION:
At baseline (BSL), subjects whose eligibility was confirmed were randomized to one of the following four treatment groups.

* 75 mg secukinumab
* 150 mg secukinumab
* 300 mg secukinumab
* Placebo At Week 16, all subjects were classified as responders (≥ 20% improvement from BSL in both tender and swollen joint counts) or non-responders.

Subjects who were randomized to a secukinumab treatment group at baseline were targeted to remain on the same dose for the entire trial.

Subjects who were randomized to placebo at baseline were re-randomized at Week 16 as follows:

Placebo non-responders received secukinumab 150 mg s.c. or 300 mg s.c. (1:1) every 4 weeks, starting after the efficacy assessments at Week 16.

Placebo responders continued to receive placebo at Week 16 and Week 20 and received secukinumab 150 mg s.c. or 300 mg s.c. (1:1) every 4 weeks, starting after the efficacy assessments at Week 24.

This was a double-blind, double-dummy, randomized treatment trial until week 52 analysis was completed and open label afterwards.

An amendment to the study protocol (after all patients were in the trial for 2-3 years) introduced changes whereby patients previously treated with secukinumab 75 mg s.c. could change to receive 150 mg s.c. or 300 mg s.c., and patients previously treated with secukinumab 150 mg s.c. could change to receive 300 mg s.c., as deemed appropriate by the investigators.

ELIGIBILITY:
Inclusion Criteria:Patients eligible for inclusion in this study have to fulfill all of the following criteria:

* Diagnosis of PsA classified by CASPAR criteria and with symptoms for at least 6 months with moderate to severe PsA who must have at Baseline ≥3 tender joints out of 78 and ≥3 swollen out of 76 (dactylitis of a digit counts as one joint each)
* Rheumatoid factor and anti-CCP antibodies negative at screening
* Diagnosis of active plaque psoriasis or nail changes consistent with psoriasis or documented history of plaque psoriasis
* Subjects with PsA should have taken NSAIDs for at least 4 weeks prior to randomization with inadequate control of symptoms or at least one dose if stopped due to intolerance to NSAIDs
* Subjects taking corticosteroids must be on a stable dose of ≤10 mg/day prednisone or equivalent for at least 2 weeks before randomization and should remain on a stable dose up to Week 24
* Subjects taking MTX (≤ 25 mg/week) are allowed to continue their medication if the dose is stable for at least 4 weeks before randomization and should remain on a stable dose up to Week 52.

Exclusion Criteria:Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

* Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician
* Subjects taking high potency opioid analgesics (e.g. methadone, hydromorphone, morphine)
* Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor
* Ongoing use of prohibited psoriasis treatments / medications (e.g., topical corticosteroids, UV therapy) at randomization. The following wash out periods need to be observed:
* Oral or topical retinoids 4 weeks
* Photochemotherapy (e.g. PUVA) 4 weeks
* Phototherapy (UVA or UVB) 2 weeks
* Topical skin treatments (except in face, scalp and genital area during screening, only corticosteroids with mild to moderate potency) 2 weeks
* Subjects who have ever received biologic immunomodulating agents except for those targeting TNFα, investigational or approved
* Previous treatment with any cell-depleting therapies including but not limited to anti-CD20, investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2013-04-14 (Actual); Primary Completion 2014-05-12 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (71):
- United States (20):
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Zephyrhills, Florida
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, League City, Texas
  - Novartis Investigative Site, Mesquite, Texas
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern East, Victoria
- Belgium (3):
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
- Canada (6):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Pointe-Claire, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (4):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Germany (8):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zerbst
- Poland (4):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Ponce, Puerto Rico
- Russia (9):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Bangkok, Thailand
- United Kingdom (11):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Cannock, Staffordshire
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Secukinumab in Patients with Psoriatic Arthritis at 52 Weeks Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):817-828. doi: 10.1007/s40744-024-00652-7. Epub 2024 Mar 6. PMID 38446397
- [Derived] McInnes IB, Mease PJ, Kivitz AJ, Nash P, Rahman P, Rech J, Conaghan PG, Kirkham B, Navarra S, Belsare AD, Delicha EM, Pricop L. Long-term efficacy and safety of secukinumab in patients with psoriatic arthritis: 5-year (end-of-study) results from the phase 3 FUTURE 2 study. Lancet Rheumatol. 2020 Apr;2(4):e227-e235. doi: 10.1016/S2665-9913(20)30036-9. PMID 38268157
- [Derived] Pournara E, Kormaksson M, Nash P, Ritchlin CT, Kirkham BW, Ligozio G, Pricop L, Ogdie A, Coates LC, Schett G, McInnes IB. Clinically relevant patient clusters identified by machine learning from the clinical development programme of secukinumab in psoriatic arthritis. RMD Open. 2021 Nov;7(3):e001845. doi: 10.1136/rmdopen-2021-001845. PMID 34795065
- [Derived] Coates LC, Wallman JK, McGonagle D, Schett GA, McInnes IB, Mease PJ, Rasouliyan L, Quebe-Fehling E, Asquith DL, Fasth AER, Pricop L, Gaillez C. Secukinumab efficacy on resolution of enthesitis in psoriatic arthritis: pooled analysis of two phase 3 studies. Arthritis Res Ther. 2019 Dec 4;21(1):266. doi: 10.1186/s13075-019-2055-z. PMID 31801620
- [Derived] Deodhar A, Gladman DD, McInnes IB, Spindeldreher S, Martin R, Pricop L, Porter B, Safi J Jr, Shete A, Bruin G. Secukinumab Immunogenicity over 52 Weeks in Patients with Psoriatic Arthritis and Ankylosing Spondylitis. J Rheumatol. 2020 Apr;47(4):539-547. doi: 10.3899/jrheum.190116. Epub 2019 Jun 15. PMID 31203228
- [Derived] Coates LC, Gladman DD, Nash P, FitzGerald O, Kavanaugh A, Kvien TK, Gossec L, Strand V, Rasouliyan L, Pricop L, Ding K, Jugl SM, Gaillez C; FUTURE 2 study group. Secukinumab provides sustained PASDAS-defined remission in psoriatic arthritis and improves health-related quality of life in patients achieving remission: 2-year results from the phase III FUTURE 2 study. Arthritis Res Ther. 2018 Dec 7;20(1):272. doi: 10.1186/s13075-018-1773-y. PMID 30526678
- [Derived] McInnes IB, Mease PJ, Schett G, Kirkham B, Strand V, Williams N, Fox T, Pricop L, Jugl SM, Gandhi KK; FUTURE 2 Study Group. Secukinumab provides rapid and sustained pain relief in psoriatic arthritis over 2 years: results from the FUTURE 2 study. Arthritis Res Ther. 2018 Jun 7;20(1):113. doi: 10.1186/s13075-018-1610-3. PMID 29880010
- [Derived] Coates LC, Mease PJ, Gossec L, Kirkham B, Sherif B, Gaillez C, Mpofu S, Jugl SM, Karyekar C, Gandhi KK. Minimal Disease Activity Among Active Psoriatic Arthritis Patients Treated With Secukinumab: 2-Year Results From a Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Phase III Study. Arthritis Care Res (Hoboken). 2018 Oct;70(10):1529-1535. doi: 10.1002/acr.23537. Epub 2018 Sep 1. PMID 29409133
- [Derived] McInnes IB, Mease PJ, Ritchlin CT, Rahman P, Gottlieb AB, Kirkham B, Kajekar R, Delicha EM, Pricop L, Mpofu S. Secukinumab sustains improvement in signs and symptoms of psoriatic arthritis: 2 year results from the phase 3 FUTURE 2 study. Rheumatology (Oxford). 2017 Nov 1;56(11):1993-2003. doi: 10.1093/rheumatology/kex301. PMID 28968735
- [Derived] McInnes IB, Mease PJ, Kirkham B, Kavanaugh A, Ritchlin CT, Rahman P, van der Heijde D, Landewe R, Conaghan PG, Gottlieb AB, Richards H, Pricop L, Ligozio G, Patekar M, Mpofu S; FUTURE 2 Study Group. Secukinumab, a human anti-interleukin-17A monoclonal antibody, in patients with psoriatic arthritis (FUTURE 2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2015 Sep 19;386(9999):1137-46. doi: 10.1016/S0140-6736(15)61134-5. Epub 2015 Jun 28. PMID 26135703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population was comprised of subjects who had passed screening assessments, complied with eligibility criteria and had provided written consent
Pre-assignment Details: At baseline, all eligible subjects were randomized via Interactive Response Technology (IRT) to one of the 4 treatment arms.
  At Week 16, Subjects on Placebo were rerandomized to receive secukinumab 150 mg s.c. or 300 mg s.c. from Week 16 (non-responder) or Week 24 (responder).
Groups:
- Secukinumab (AIN457) 75 mg s.c.: Secukinumab 75 mg at BSL, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4 until up to Week 260. After a protocol amendment (introduced in open label phase > 2 years post randomization) patients could be changed to 150 mg s.c. or 300 mg s.c
- Secukinumab (AIN457) 150 mg s.c.: Secukinumab 150 mg at BSL, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4 until up to Week 260. After a protocol amendment (introduced in open label phase > 2 years post randomization) patients could be changed to 300 mg s.c
- Secukinumab (AIN457) 300 mg s.c.: Secukinumab 300 mg at BSL, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4 until up to Week 260.
- Placebo - AIN457 150 mg: Placebo - rerandomized to AIN457 150 mg starting at Week 16 (non-responder) or Week 24 (responder). After a protocol amendment (introduced in open label phase > 2 years post randomization) patients could be changed to 300 mg s.c
- Placebo - AIN457 300 mg: Placebo - rerandomized to AIN457 300 mg starting at Week 16 (non-responder) or Week 24 (responder).
- Placebo - Not Rerandomized: Placebo - not rerandomized (subjects discontinued prior to rerandomization scheduled for week 16)
Period: Up to Week 24 (Primary Analysis)
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Placebo - Not Rerandomized
Started | 99 | 100 | 100 | 43 | 45 | 10
Completed | 93 | 95 | 97 | 43 | 45 | 0
Not Completed | 6 | 5 | 3 | 0 | 0 | 10
Not completed — Subject/guardian decision | 1 | 1 | 1 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 3 | 0 | 2 | 0 | 0 | 4
Period: Week 24 to Week 260
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Placebo - Not Rerandomized
Started | 93 | 95 | 97 | 43 | 45 | 0
Completed | 59 | 65 | 64 | 29 | 31 | 0
Not Completed | 34 | 30 | 33 | 14 | 14 | 0
Not completed — Lack of Efficacy | 15 | 7 | 7 | 3 | 4 | 0
Not completed — Subject/guardian decision | 12 | 10 | 9 | 5 | 5 | 0
Not completed — Physician Decision | 1 | 2 | 4 | 2 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Noncompliance with study treatment | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 3 | 0 | 2 | 0
Not completed — Adverse Event | 4 | 8 | 8 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Placebo - Not Rerandomized | Total
Number analyzed (Participants) | 99 | 100 | 100 | 43 | 45 | 10 | 397
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 93 | 94 | 90 | 36 | 43 | 8 | 364
  >=65 years | 6 | 6 | 10 | 7 | 2 | 2 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 49 | 24 | 29 | 6 | 205
  Male | 47 | 55 | 51 | 19 | 16 | 4 | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Asian | 5 | 6 | 2 | 0 | 1 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 90 | 90 | 96 | 42 | 43 | 9 | 370
  More than one race | 2 | 1 | 1 | 1 | 1 | 1 | 7
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving American College of Rheumatology 20 (ACR20) Response Criteria
Description: ACR20 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
  For subjects with early escape at Week 16 or had missing values at Week 24 or discontinued prior to Week 24, their ACR20 was set to nonresponse at Week 24. This applied for all treatment regimens in order to minimize bias. The Placebo arm was analyzed as one group, irrespective of the re-randomization, as assessments made under the re-randomized active treatment were not included in this analysis.
Time Frame: Week 24
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo s.c.: Placebo at BSL, Weeks 1, 2, 3 and 4, followed by placebo dosing every four weeks starting at Week 4 until up to Week 12 (non-responder) or Week 20 (responder) followed by re-randomization to AIN 150 mg s.c. or AIN 300 mg s.c. (starting from Week 16 or 24). After a protocol amendment (introduced in open label phase > 2 years post randomization) patients re-randomized to 150 mg s.c. could be changed to 300 mg s.c. Treatment could continue up to Week 260.
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 99 | 100 | 100 | 98
Participants | 29 | 51 | 54 | 15
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0200, Regression, Logistic; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.14 to 4.73]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p < 0001, Regression, Logistic; Odds Ratio (OR) = 6.52, 95% CI 2-sided [3.25 to 13.08]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 6.81, 95% CI 2-sided [3.42 to 13.56]

2. Secondary Outcome: Number of Participants Achieving a PASI75 Response in the Subgroup of Subjects Who Have ≥3% Skin Involvement With Psoriasis
Description: PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI 75 response was defined as participants achieving >= 75% improvement from baseline. For subjects with early escape at Week 16 or had missing values at Week 24 or discontinued prior to Week 24, their value was set to nonresponse at Week 24. This applied for all treatment regimens in order to minimize bias.
Time Frame: Week 24
Population: Psoriasis Subset (≥3% skin involvement with psoriasis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 50 | 58 | 41 | 43
Participants | 14 | 28 | 26 | 7
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.1650, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.74 to 5.81]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 5.70, 95% CI 2-sided [2.12 to 15.34]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 9.48, 95% CI 2-sided [3.33 to 27.00]

3. Secondary Outcome: Number of Participants Achieving a PASI90 Response in the Subgroup of Subjects Who Have ≥3% Skin Involvement With Psoriasis
Description: PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI 90 response was defined as participants achieving >= 90% improvement from baseline. For subjects with early escape at Week 16 or had missing values at Week 24 or discontinued prior to Week 24, their value was set to nonresponse at Week 24. This applied for all treatment regimens in order to minimize bias.
Time Frame: Week 24
Population: Psoriasis Subset (≥3% skin involvement with psoriasis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 50 | 58 | 41 | 43
Participants | 6 | 19 | 20 | 4
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.6421, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.36 to 5.36]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0029, Regression, Logistic; Odds Ratio (OR) = 6.36, 95% CI 2-sided [1.89 to 21.47]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 10.74, 95% CI 2-sided [3.13 to 36.84]

4. Secondary Outcome: Change From Baseline in DAS28-CRP
Description: The DAS28 is a measure of disease activity based on Swollen and Tender Joint Counts, ESR or CRP and the Patient Global Assessment. A DAS28 score > 5.1 implies active disease, ≤ 3.2 low disease activity, and < 2.6 remission. The score can range from 0 - 9.4. The data collected after the patient switched to secukinumab were treated as missing for placebo patients and were analyzed using a mixed-effects repeated measures model. For secukinumab patients, the actual values were used in the analysis.
  The Placebo arm was analyzed as one group, irrespective of the re-randomization, as assessments made under the re-randomized active treatment were not included in this analysis.
Time Frame: Baseline, Week 24
Population: Full Analysis Set, including only participants with measurements at baseline and Week 24. Participants in the Placebo arm who switched to Secukinumab prior to Week 24 were treated as missing.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 87 | 91 | 93 | 32
score on a scale | -1.12 (0.111) | -1.58 (0.109) | -1.61 (0.110) | -0.96 (0.149)
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.3763, Mixed Models Analysis; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.53 to 0.20]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Mean Difference (Net) = -0.62, 95% CI 2-sided [-0.98 to -0.26]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.02 to -0.29]

5. Secondary Outcome: Change From Baseline in SF36-Physical Component Score
Description: The SF-36 is an instrument to measure health-related quality of life among healthy patients and patients with acute and chronic conditions.
  Score range is from 0 (no problems) to 100 (unable to perform the activity). SF-36 is a 36 item questionnaire which measures Quality of Life across eight domains, which are both physically and emotionally based. Two overall summary scores, the Physical Component Summary (PCS) and Mental Component Summary (MCS) can be computed. In this study, SF-36 PCS was used.
  The Placebo arm was analyzed as one group, irrespective of the re-randomization, as assessments made under the re-randomized active treatment were not included in this analysis.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 91 | 96 | 96 | 33
Score on a scale | 4.38 (0.750) | 6.39 (0.734) | 7.25 (0.740) | 1.95 (0.974)
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0482, Mixed Models Analysis; Mean Difference (Net) = 2.42, 95% CI 2-sided [0.02 to 4.83]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = 4.44, 95% CI 2-sided [2.05 to 6.83]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 5.30, 95% CI 2-sided [2.91 to 7.69]

6. Secondary Outcome: Change From Baseline in Stanford Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement. The Placebo arm was analyzed as one group, irrespective of the re-randomization, as assessments made under the re-randomized active treatment were not included in this analysis.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 89 | 95 | 95 | 33
Scores on a scale | -0.32 (0.050) | -0.48 (0.049) | -0.56 (0.050) | -0.31 (0.060)
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.9195, Mixed Models Analysis; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.16 to 0.15]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0278, Mixed Models Analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.32 to -0.02]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0013, Mixed Models Analysis; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.40 to -0.10]

7. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 50 (ACR50) Response Criteria
Description: ACR20 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 50% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). For subjects with early escape at Week 16 or had missing values at Week 24 or discontinued prior to Week 24, their ACR20 was set to nonresponse at Week 24. This applied for all treatment regimens in order to minimize bias. The Placebo arm was analyzed as one group, irrespective of the re-randomization, as assessments made under the re-randomized active treatment were not included in this analysis.
Time Frame: Week 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 99 | 100 | 100 | 98
Participants | 18 | 35 | 35 | 7
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0245, Regression, Logistic; Odds Ratio (OR) = 2.91, 95% CI 2-sided [1.15 to 7.36]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 7.54, 95% CI 2-sided [3.11 to 18.25]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 7.15, 95% CI 2-sided [2.97 to 17.22]

8. Secondary Outcome: Number of Participants With Dactylitis in the Subset of Subjects Who Had Dactylitis at Baseline
Description: Resolution of dactylitis was evaluated in the subset of patients who had disease activity at baseline. In this analysis, a lower percentage is desirable and resolution is defined as complete absence of the symptom. For subjects with early escape at Week 16 or had missing values at Week 24 or discontinued prior to Week 24, their assessment was set to nonresponse at Week 24 (presence of dactylitis). This applied for all treatment regimens in order to minimize bias. The Placebo arm was analyzed as one group, irrespective of the re-randomization, as assessments made under the re-randomized active treatment were not included in this analysis.
Time Frame: Week 24
Population: Dactylitis Subset (participants with dactylitis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 33 | 32 | 46 | 27
Participants | 23 | 16 | 20 | 23
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.3149, Regression, Logistic; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.13 to 1.91]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0056, Regression, Logistic; Odds Ratio (OR) = 0.16, 95% CI 2-sided [0.04 to 0.58]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 0.14, 95% CI 2-sided [0.04 to 0.50]

9. Secondary Outcome: Number of Participants With Enthesitis in the Subset of Subjects Who Had Enthesitis at Baseline
Description: Resolution of enthesitis was evaluated in the subset of patients who had disease activity at baseline. In this analysis, a lower percentage is desirable and resolution is defined as complete absence of the symptom. For subjects with early escape at Week 16 or had missing values at Week 24 or discontinued prior to Week 24, their assessment was set to nonresponse at Week 24 (presence of enthesitis). This applied for all treatment regimens in order to minimize bias. The Placebo arm was analyzed as one group, irrespective of the re-randomization, as assessments made under the re-randomized active treatment were not included in this analysis.
Time Frame: Week 24
Population: Enthesitis Subset (participants with enthesitis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab (AIN457) 75 mg s.c. | Secukinumab (AIN457) 150 mg s.c. | Secukinumab (AIN457) 300 mg s.c. | Placebo s.c.
Number analyzed (Participants) | 68 | 64 | 56 | 65
Participants | 46 | 37 | 29 | 51
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 75 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.1678, Regression, Logistic; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.26 to 1.26]
Statistical Analysis 2: Comparison: Secukinumab (AIN457) 150 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0108, Regression, Logistic; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.17 to 0.79]
Statistical Analysis 3: Comparison: Secukinumab (AIN457) 300 mg s.c. vs Placebo s.c; Test type: Superiority; p = 0.0025, Regression, Logistic; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.13 to 0.65]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until Last Patient Last Visit (LPLV), up to a maximum of 5 years.
Description: Patients randomized to Placebo at Baseline are reported under Placebo for AEs starting before switching to Secukinumab (non-responder Week 16 / responder Week 24) and under the respective Secukinumab arm for AEs starting after switching to Secukinumab. Patients who, following the protocol amendment, switched to a higher dose are reporteed under the arm (dose) where the AE occurred.
Groups:
- Any AIN457 75 mg: Any AIN457 75 mg
- Any AIN457 150 mg: Any AIN457 150 mg
- Any AIN457 300 mg: Any AIN457 300 mg
- Placebo: Placebo
Arm/Group | Any AIN457 75 mg | Any AIN457 150 mg | Any AIN457 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 1/193 | 0/251 | 0/98
Serious Adverse Events (participants affected / at risk) | 17/99 | 28/193 | 42/251 | 3/98
Other Adverse Events (participants affected / at risk) | 63/99 | 132/193 | 171/251 | 39/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=99) | Any AIN457 150 mg (N=193) | Any AIN457 300 mg (N=251) | Placebo (N=98)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced transiently (Eye disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 2 | 0
Periorbital abscess (Infections and infestations) | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Dependence (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pregnancy of partner (Social circumstances) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Vasculitis necrotising (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=99) | Any AIN457 150 mg (N=193) | Any AIN457 300 mg (N=251) | Placebo (N=98)
Diarrhoea (Gastrointestinal disorders) | 11 | 19 | 23 | 3
Nausea (Gastrointestinal disorders) | 7 | 12 | 14 | 4
Fatigue (General disorders) | 5 | 6 | 11 | 2
Oedema peripheral (General disorders) | 5 | 3 | 4 | 0
Bronchitis (Infections and infestations) | 7 | 13 | 19 | 2
Influenza (Infections and infestations) | 3 | 10 | 14 | 0
Nasopharyngitis (Infections and infestations) | 23 | 41 | 47 | 8
Oral herpes (Infections and infestations) | 5 | 2 | 8 | 2
Pharyngitis (Infections and infestations) | 1 | 6 | 15 | 0
Respiratory tract infection (Infections and infestations) | 5 | 5 | 7 | 0
Rhinitis (Infections and infestations) | 5 | 6 | 9 | 0
Sinusitis (Infections and infestations) | 6 | 16 | 30 | 1
Upper respiratory tract infection (Infections and infestations) | 23 | 40 | 58 | 7
Urinary tract infection (Infections and infestations) | 8 | 16 | 19 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 24 | 25 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 11 | 21 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 5 | 7 | 8 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 12 | 12 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 11 | 3
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 12 | 24 | 23 | 2
Headache (Nervous system disorders) | 6 | 16 | 18 | 5
Depression (Psychiatric disorders) | 5 | 4 | 14 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 13 | 12 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 7 | 14 | 17 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 8 | 13 | 3
Hypertension (Vascular disorders) | 6 | 14 | 23 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.